CLINICAL TRIAL: NCT02907138
Title: Medical Yoga for Patients With Stress-related Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Larsson (Other Government)
Responsible Party: Sponsor-Investigator, Maria Larsson, Assoc. professor, Research and Development director, Vastra Gotaland Region
Organization: Vastra Gotaland Region (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VGFOUGSB-602221
Record Dates: First submitted 2016-09-09; First posted 2016-09-20 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Stress-related Illness/Anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Therapeutics; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Medical Yoga (Experimental): Medical Yoga Group therapy for eight weeks, 60 minutes per week, with the guidance of a physical therapist.
  Interventions: Other: Medical Yoga
- Treatment as Usual (physical therapy) (Active Comparator): Treatment as Usual provided by physical therapist
  Interventions: Other: Treatment as Usual (physical therapy)

INTERVENTIONS:
Other: Medical Yoga
  Arms: Medical Yoga
Other: Treatment as Usual (physical therapy)
  Arms: Treatment as Usual (physical therapy)

SUMMARY:
The purpose of this study is to compare the effect of Medical Yoga as a group treatment, to conventional treatment provided by a physical therapist, for people with perceived stress-related symptoms.

Forty people are to be randomized to either:

1. Intervention Group - Medical Yoga, group treatment for eight weeks, 60 minutes per week, with the guidance of a physical therapist.

   or
2. Control - treatment as usual (TAU) in physical therapy.

ELIGIBILITY:
Inclusion Criteria:

* Perceived stress and anxiety, which could be expressed as for example as tension in the neck and shoulders, insomnia, anxiety and headaches.

Exclusion Criteria:

* Do not understand Swedish (as group instructions need to be understood),
* Pregnancy,
* Psychotic symptoms,
* Ongoing or physical therapy treatment the last three months,
* Previously participated in Medical Yoga group.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-09; Primary Completion 2019-02-15 (Actual); Study Completion 2019-03-04 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS) | baseline, follow-up at approx 8 weeks after first treatment session, follow-up at approx 20 weeks after first treatment session
  Outcome will be measured as change between baseline and follow-ups and between follow-ups. Total score will also be analysed between groups at follow-up(s).

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | baseline, follow-up at approx 8 weeks after first treatment session, follow-up at approx 20 weeks after first treatment session
Health-related quality of Life; EQ5D | baseline, follow-up at approx 8 weeks after first treatment session, follow-up at approx 20 weeks after first treatment session
Thorax excursion: Measured in centimeters with tape measure, chest size at the level of processus xiphoideus, the difference between the maximum inhalation and exhalation is registered | baseline, follow-up at approx 8 weeks after first treatment session, follow-up at approx 20 weeks after first treatment session
Health-related quality of Life; EQ-VAS | baseline, follow-up at approx 8 weeks after first treatment session, follow-up at approx 20 weeks after first treatment session

CONTACTS AND LOCATIONS:
Locations (1):
- Narhalsan Gibraltar rehabmottagning, Gothenburg, Sweden

REFERENCES:
- [Derived] Bellfjord M, Grimby-Ekman A, Larsson MEH. MediYoga compared to physiotherapy treatment as usual for patients with stress-related symptoms in primary care rehabilitation: A randomized controlled trial. PLoS One. 2024 Jun 13;19(6):e0300756. doi: 10.1371/journal.pone.0300756. eCollection 2024. PMID 38870156